CLINICAL TRIAL: NCT01528748
Title: Clinical Trial of CBASP for Individuals With Co-occurring Chronic Depression and Alcohol Dependence
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jennifer Kim Penberthy, Associate Professor, School of Medicine, University of Virginia
Other Study IDs: 15599
Record Dates: First submitted 2012-02-04; First posted 2012-02-08 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Depressive Disorder; Major Depressive Disorder; Dysthymic Disorder; Alcohol-Related Disorders; Alcoholism
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Dysthymic Disorder; Alcohol-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronically Depressed, Alcohol Dependent: Participants who have been formally diagnosed with a clinical diagnosis of Chronic Depression and Alcohol Dependence.
  Interventions: Behavioral: Cognitive Behavioral Analysis System of Psychotherapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Analysis System of Psychotherapy — Cognitive Behavioral Analysis System of Psychotherapy (CBASP) is a behavioral intervention that addresses the unique behavioral characteristics of chronically depressed individuals, most of which are highly relevant for alcoholics as well. CBASP has a structured, individualized, and collaborative (patient and clinician) design. The intervention emphasizes teaching effective coping strategies and employing motivational, cognitive, behavioral, and interpersonal techniques. Individual therapy (1 hour) sessions occur on a weekly basis for a total of 20 sessions over a period of 21 weeks.
  Other Names: CBASP

SUMMARY:
This study examines the effectiveness of Cognitive Behavioral Analysis System of Psychotherapy (CBASP) in reducing both alcohol consumption and depressive symptoms in adults who are chronically depressed and alcohol dependent.

DETAILED DESCRIPTION:
This study examines the effectiveness of Cognitive Behavioral Analysis System of Psychotherapy (CBASP) in reducing both alcohol consumption and depressive symptoms in adults who are chronically depressed and alcohol dependent. Participants will receive a 20-session course of CBASP psychotherapy over a period of 21 weeks and will be assessed for severity of pretreatment psychological abuse and trauma as well as pre and posttreatment interpersonal functioning. Two primary hypotheses are to be tested: 1) demonstrate that CBASP is effective in reducing depressive symptoms (Hamilton Rating Scale for Depression-24 ratings) and alcohol consumption (drinks per drinking day) in this chronically depressed alcohol dependent cohort when posttreatment ratings are compared to pretreatment levels; and 2) demonstrate that acquisition of feeling safe with the therapist and acquisition of the ability to perceive the interpersonal consequences of one's behavior will significantly increase from pre to posttreatment levels and will be associated with reductions in drinking and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a current major depressive disorder (e.g., Major Depression, Dysthymic Disorder) for a minimum of two years
* Clinical diagnosis of alcohol dependence during the last thirty days
* Interest in changing one's drinking and alleviating depressive symptoms

Exclusion Criteria:

* Please call study site for additional information

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited via a community sample.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Depression Rating | Baseline and 20 weeks
  Change in depression rating scale over time.
Drinking behavior | Baseline and 20 weeks
  Change in number of drinks consumed per day over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K. Penberthy, Ph.D., Principal Investigator — University of Virginia, School of Medicine, Department of Psychiatry & Neurobehavioral Sciences
Locations (1):
- University of Virginia Center for Addiction Research & Education (UVa CARE), Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCullough JP Jr. Treatment for chronic depression using Cognitive Behavioral Analysis System of Psychotherapy (CBASP). J Clin Psychol. 2003 Aug;59(8):833-46. doi: 10.1002/jclp.10176. PMID 12858425
- [Background] McCullough, Jr., JP. (2001). Skills Training Manual for Diagnosis and Treating Chronic Depression: Cognitive Behavioral Analysis System of Psychotherapy (CBASP). New York: Guilford Press.